CLINICAL TRIAL: NCT01599143
Title: Identifying Therapeutic Factors in an 8-Week (30 Hour) Mindfulness-Based Stress Reduction (MBSR) Program
Acronym: mbsr
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: North York General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Katalin Margittai, Assistant Professor of Psychiatry, University of Toronto, North York General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NYGH REB # 09-0041
Record Dates: First submitted 2012-04-30; First posted 2012-05-15 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Cancer; Diabetes; Hypertension
Keywords: Mindfulness; Pain Disorder (Chronic physical or mental health complaints:; Fibromyalgia; Migraines; Back Pain; etc); Anxiety Disorder/Anxiety State
MeSH Terms: conditions — Neoplasms; Diabetes Mellitus; Hypertension; Somatoform Disorders; Fibromyalgia; Migraine Disorders; Back Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mindfulness-based Stress Reduction group (Experimental): All eligible participants attend a 3-hour weekly session, for 8 consecutive weeks, to learn meditation and simple Hatha Yoga techniques, and incorporate them into their daily lives.
  Interventions: Behavioral: Teaching Mindfulness-based Stress Reduction strategies

INTERVENTIONS:
Behavioral: Teaching Mindfulness-based Stress Reduction strategies — Daily meditation, Hatha yoga,and cognitive restructuring
  Other Names: MBSR

SUMMARY:
Since it's introduction in 1979 at the University of Massachusetts Medical Center by Dr. Jon Kabat-Zinn, Mindfulness-Based Stress Reduction (MBSR) has become a respected adjunct to conventional treatment for patients suffering from many diverse chronic ailments. Three decades of research have documented it's benefits, but few papers have focused on identifying which particular aspect of MBSR directly correlates with it's degree of therapeutic efficacy. This study will use 7 well validated questionnaires to compare participants responses prior to, and following completion of an eight-week MBSR program at the North York General Hospital, as well as follow-up results at 1 month and 1 year post completion of the MBSR group.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* suffer from a chronic health problem
* referred by their physician

Exclusion Criteria:

* acute illness (physical or psychiatric)
* suicidal
* problem use of alcohol or other substances
* inability to do one hour of daily homework
* inability to attend all 8 sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2009-01; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
PSS-10 | baseline, 8 weeks and follow-ups at 1 month and 1 year
  Patients' Stress Scores on the PSS-10 are used to assess self-reported perceptions of stress at baseline, at 8 weeks when the intervention ends, and again at one month and one year follow-up (to see if any change is sustained).

SECONDARY OUTCOMES:
Toronto Mindfulness Scale (TMS) | Baseline, 8 weeks and follow up at 1 month and 1 year
  Measure of patients' self-reported capacity for detached curiosity / decentering (aspects of mindfulness), prior to intervention, at the end of the intervention (8 weeks), and at short-term (one month)and long-term (one year) follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Katalin J Margittai, MD, Principal Investigator — North York General Hospital